CLINICAL TRIAL: NCT01423292
Title: Ultrasound Guided Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia After Laparoscopic Colonic Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji Won Park, Center for Colorectal Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCCTS-11-557
Record Dates: First submitted 2011-08-18; First posted 2011-08-25 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Laparoscopic Colecctomy
MeSH Terms: interventions — Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- an odd numbered patients (Active Comparator): TAP block with local anesthetics
  Interventions: Procedure: Ultrasound Guided Transversus Abdominis Plane (TAP) Block; Drug: bupivacaine
- an even numbered patients (Placebo Comparator): TAP block without local anesthetics
  Interventions: Procedure: Ultrasound Guided Transversus Abdominis Plane (TAP) Block; Drug: Placebo

INTERVENTIONS:
Procedure: Ultrasound Guided Transversus Abdominis Plane (TAP) Block — Ultrasound Guided Transversus Abdominis Plane (TAP) Block
Drug: bupivacaine — 0.25 bupivacaine 30ml (15ml on each side)
  Arms: an odd numbered patients
Drug: Placebo — placebo
  Arms: an even numbered patients

SUMMARY:
The purpose of this study is to determine whether the transversus abdominis plane (TAP) blocks are effective in postoperative pain control of adult patients undergoing laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

* aged 20~80
* undergoing laparoscopic colectomy

Exclusion Criteria:

* allergic history to local anesthesitcs
* tolerance to opioid
* cannot use IV-PCA
* previous abdominal surgery
* intestinal obstruction
* emergency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
pain score during cough | 24hr after TAP block
  pain score during cough at 24 hours after TAP block (using visual analog scale)

SECONDARY OUTCOMES:
pain score during bed rest and ambulation at ward, dosage of used opioid, nausea score, sedation score, days of hospitalization, start day of diet, reinsertion rate of urinary catheter, satisfaction measurement of pain control, life of quality | 24hr, 48hr, 72hr after TAP block

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea